CLINICAL TRIAL: NCT00511043
Title: Phase II Open Label Study of PTK787/ZK222584 in Adults Patients With Refractory or Relapsed Diffuse Large Cell Lymphoma
Brief Title: PTK787 in Refractory or Relapsed Diffuse Large Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer stopped drug development
Sponsor: David Rizzieri, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Division of Cellular Therapy, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008648; CPTK787AUS39; 7416 (Other: Legacy Duke IRB number)
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-11

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: PTK787; DLCL; Diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All pts (Experimental): PTK787
  Interventions: Drug: PTK787

INTERVENTIONS:
Drug: PTK787 — PTK787 - 1250mg p.o. daily. Initial dose of 750mg p.o daily starting on day 1 and increased weekly to an intermediate dose of 1000 mg and then a target dose of 1250mg unless a grade ≥ 2 toxicity. Patients who tolerate the study target dose of 1250mg will remain on that dose until study completion at 12 months or until disease progression, unacceptable toxicity, withdrawal of consent or patient non-compliance with the protocol requirement.
  Other Names: Vatalanib; ZK 222584; PTK787/ZK 222584

SUMMARY:
This is a phase II open label study to assess the efficacy and safety of PTK787/ZK222584 in adults with relapsed or refractory diffuse large cell lymphoma (DLCL). All subjects will receive PTK787/ZK222584. Subjects who tolerate the study target dose of 1250mg will remain on that dose until study completion at 12 months or until disease progression, unacceptable toxicity, withdrawal of consent or non-compliance with the protocol requirement.

DETAILED DESCRIPTION:
In order for tumors to grow and spread to other parts of the body, they need to have a growing blood supply. Tumor cells have been shown to produce substances that stimulate the abnormal growth of new blood vessels that allow the tumor to grow. In adults, blood vessel cells normally divide very rapidly. It is thought that PTK787/ZK222584 may interfere with the growth of new blood vessels. A drug that interferes with the growth of new blood vessels might stop tumor growth, and possibly shrink the tumor by keeping it from receiving nutrients and oxygen supplied by the blood vessels. Since normal blood vessel cells divide very rapidly, it might be possible to stop tumor growth without harming normal tissues.

The purpose of this study is to find out if an investigational drug, PTK787/ZK 222584 is safe and effective in treating relapsed or refractory diffuse large cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLCL (de novo or transformed).
* Measurable/evaluable disease by radiographs, physical exam or bone marrow involvement.
* Refractory disease, induction chemotherapy failure or relapsed disease.
* Age ≥ 18 years old
* Performance Status:KPS ≥ 70
* Laboratory tests as specified by the protocol.
* Written informed consent

Exclusion Criteria:

* History of known central nervous system disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis).
* History of another primary malignancy ≤ 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin
* Prior chemotherapy ≤ 3 weeks prior to registration. There is no limit to the number of prior chemotherapy regimens.
* Prior allogeneic transplant if >2.5% donor cells remain by engraftment studies (prior autologous transplant is allowed)
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration.
* Prior full field (total organ site) radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to registration.
* Major surgery (i.e., laparotomy) ≤ 4 weeks prior to registration. Minor surgery ≤ 2 weeks prior to registration.
* Patients who have received investigational drugs ≤ 4 weeks prior to registration and/or registration
* Prior therapy with anti-VEGF targeted agents
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* QTc > 450 (male) or > 470 (female). Patients with congenital or acquired prolonged QTc syndrome
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control.
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
  * Unstable angina pectoris
  * Symptomatic congestive heart failure
  * Myocardial infarction ≤ 6 months prior to registration
  * Serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes
  * Severe active or uncontrolled infection
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease with documented nephritic or nephrotic syndrome.
* Acute or chronic liver disease
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK222584
* Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if he/she feels that 1) a potential drug interaction between PTK787/ZK 222584 and anti-HIV medications that could influence the efficacy of the anti-HIV medication, or 2) it may place the patient at risk due to the pharmacologic activity of PTK787/ZK 222584.
* Patients who are taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system.
* Patients unwilling to or unable to comply with the protocol
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response | approximately 1 year

SECONDARY OUTCOMES:
Safety | 30 days post last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - South Carolina Oncology Associates, Columbia, North Carolina
  - Duke University Medical Center, Durham, North Carolina